CLINICAL TRIAL: NCT04046588
Title: The Difference in Heat Transport Characteristics of the Heart and Lung Meridians: a Comparative Study of COPD Patients and Healthy Subjects
Brief Title: The Difference in Heat Transport Characteristics of the Heart and Lung Meridians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019ZY006-MERIDIAN
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: meridians; acupuncture; chronic obstructive pulmonary disease; meridian phenomenon; infrared thermography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Moxibustion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COPD group (Other): This group will include 40 patients with chronic obstructive pulmonary disease (COPD).
  Interventions: Diagnostic Test: Infrared thermography
- Healthy control group (Other): This group will include 40 healthy volunteers.
  Interventions: Diagnostic Test: Infrared thermography
- Healthy intervention group (Experimental): This study will include 40 healthy adults. Two sessions of moxibustion intervention will be performed in the Heart meridian and Lung meridian successively.
  Interventions: Procedure: Moxibustion

INTERVENTIONS:
Diagnostic Test: Infrared thermography — A thermal imager (NEC InfRec R450, Avio Infrared Technologies Co., Ltd., Tokyo) will be used to record thermal images. The temperature of corresponding sites on the Heart and Lung meridians will be analyzed.
  Arms: COPD group; Healthy control group
Procedure: Moxibustion — Two sessions of moxibustion intervention will be performed in the Heart meridian and Lung meridian, respectivey. During moxibustion, the temperature change of relevant sites in the Heart and Lung meridians will be measured by infrared thermal imaging.
  1. Intervention in the Heart meridian: moxibustion will be performed above the acupoint HT3 of the Heart meridian
  2. Intervention in the Lung meridian: moxibustion will be performed above the acupoint LU5 of the Lung meridian.
  Other Names: Infrared thermography
  Arms: Healthy intervention group

SUMMARY:
Although some important progresses were made in the field of the meridian research, no breakthroughs have been achieved. Besides,there are some problems in meridian researches. Particularly, previous research of meridian phenomenon involved lots of subjective elements and outcomes.Researches that use modern scientific techniques to investigate the biological characteristics of meridian phenomenon are urgently needed. Therefore, this study is designed to assess the heat transport characteristics of meridian phenomenon for the Heart and Lung meridians by using infrared thermography. Thus, the biological characteristics of meridian phenomenon could be presented objectively in a scientific methodology.

DETAILED DESCRIPTION:
This study will include 40 patients with chronic obstructive pulmonary disease (COPD) and 80 healthy adults. Infrared thermal imaging(ITI) examination will be adopted to assess the heat transport characteristics of the Heart and Lung meridians and investigate the specificity for the meridian-visceral correlation and site-to-site correlation between two specific meridians.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for COPD

1. Patients should meet the above diagnostic criteria, and the severity of COPD is in the stage of GOLD 2 or 3 based on pulmonary function testing;
2. COPD patients in the stable phase, who present with mild symptoms of cough, expectoration and short breath;
3. 35 ≤ age ≤75 years, male or female;
4. Patients have clear consciousness and could communicate with others normally;
5. Patients could understand the full study protocol and have high adherence.Written informed consent is signed by themselves or their lineal kin.

Inclusion criteria for health volunteers

1. Healthy volunteers who could provide a recent medical examination report to confirm they have not any cardiovascular, respiratory, digestive, urinary, hematological, endocrine and neurological disease;
2. 35 ≤ age ≤75 years, male or female;
3. Participants have clear consciousness and could communicate with others normally;
4. Participants could understand the full study protocol and have high adherence .Written informed consent is signed by themselves or their lineal kin.

Exclusion Criteria:

Exclusion criteria for COPD

1. Patients who fail to meet the diagnostic criteria for COPD, or COPD patients in the phase of acute exacerbation;
2. Patients have the following complications, which includes pneumonia, bronchial asthma, bronchiectasis, active tuberculosis, pneumothorax, chest trauma, tumors of the lung or thorax, and other confirmed respiratory diseases;
3. Patients have concomitant conditions of heart diseases, such as chronic stable angina pectoris (CSAP);
4. Patients have serious concomitant conditions and fail to treat them effectively, such as diseases of the digestive, urinary, respiratory, hematological, and nervous system;
5. Patients have mental illness, severe depression, alcohol dependence or history of drug abuse;
6. Pregnant or lactating patients; Patients are participating in other trials.

Exclusion criteria of health volunteers

1. Participants have mental illness, severe depression, alcohol dependence or history of drug abuse;
2. Pregnant or lactating participants ;
3. Participants are participating in other trials.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Temperature change of relevant sites | Baseline, 15 minutes during moxibustion, 5 minutes after stopping moxibustion
  Infrared thermal imaging is used to record baseline temperature and the temperature change of corresponding sites along the Heart and Lung meridians.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Ph.D, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai W, Chen AW, Ding L, Shen WD. Thermal Effects of Acupuncture by the Infrared Thermography Test in Patients With Tinnitus. J Acupunct Meridian Stud. 2019 Aug;12(4):131-135. doi: 10.1016/j.jams.2019.05.002. Epub 2019 Jun 27. PMID 31254681
- [Background] Alvarez-Prats D, Carvajal-Fernandez O, Valera Garrido F, Pecos-Martin D, Garcia-Godino A, Santafe MM, Medina-Mirapeix F. Acupuncture Points and Perforating Cutaneous Vessels Identified Using Infrared Thermography: A Cross-Sectional Pilot Study. Evid Based Complement Alternat Med. 2019 Mar 21;2019:7126439. doi: 10.1155/2019/7126439. eCollection 2019. PMID 31015854
- [Background] Lin M, Wei H, Zhao L, Zhao J, Cheng K, Deng H, Shen X, Zhang H. [Review on infrared temperature characteristics of acupoints in recent 10 years]. Zhongguo Zhen Jiu. 2017 Apr 12;37(4):453-456. doi: 10.13703/j.0255-2930.2017.04.028. Chinese. PMID 29231602
- [Background] Fu Y, Ni JX, Marmori F, Zhu Q, Tan C, Zhao JP. Infrared thermal imaging-based research on the intermediate structures of the lung and large intestine exterior-interior relationship in asthma patients. Chin J Integr Med. 2016 Nov;22(11):855-860. doi: 10.1007/s11655-016-2102-4. Epub 2016 Jun 9. PMID 27286712
- [Background] de Souza RC, Pansini M, Arruda G, Valente C, Brioschi ML. Laser acupuncture causes thermal changes in small intestine meridian pathway. Lasers Med Sci. 2016 Nov;31(8):1645-1649. doi: 10.1007/s10103-016-2032-6. Epub 2016 Aug 5. PMID 27495129
- [Background] Yang H, Park H, Lim C, Park S, Lee K. Infrared thermal imaging in patients with medial collateral ligament injury of the knee - a retrospective study. J Pharmacopuncture. 2014 Dec;17(4):50-4. doi: 10.3831/KPI.2014.17.036. PMID 25780719
- [Background] Zheng J, Zhao Y, Wang Y, Hu S, Lu P, Shen X. The infrared radiation temperature characteristic of acupoints of mammary gland hyperplasia patients. Evid Based Complement Alternat Med. 2013;2013:567987. doi: 10.1155/2013/567987. Epub 2013 Nov 14. PMID 24327822
- [Background] Kang J, Lee N, Ahn Y, Lee H. Study on improving blood flow with Korean red ginseng substances using digital infrared thermal imaging and Doppler sonography: randomized, double blind, placebo-controlled clinical trial with parallel design. J Tradit Chin Med. 2013 Feb;33(1):39-45. doi: 10.1016/s0254-6272(13)60098-9. PMID 23596810
- [Derived] Li X, Jiang Y, Hu H, Zhang Y, Lou J, He X, Sun J, Wu Y, Fang J, Shao X, Fang J. The difference in heat transport characteristics of the heart and lung meridians: A comparative study of COPD patients and healthy subjects. Medicine (Baltimore). 2021 Feb 5;100(5):e23804. doi: 10.1097/MD.0000000000023804. PMID 33592838